CLINICAL TRIAL: NCT00580190
Title: A Phase I, Randomized, Placebo Controlled, Parallel Group, Single Dose Study To Evaluate The Effects Of PF-00572778 And Alprazolam On A Naloxone Challenge In Healthy Adult Subjects
Brief Title: Evaluation Of PF-00572778 And Alprazolam On Naloxone Challenge In Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Date of termination was Feb. 7, 2008. Reasons of termination were due to elevation of liver function tests and long elimination half-life of the compound.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A8821006
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: alprazolam
- 2 (Placebo Comparator)
  Interventions: Other: Placebo
- 3 (Experimental)
  Interventions: Drug: PF-00572778

INTERVENTIONS:
Drug: alprazolam — tablet, 0.5 mg, single dose, only on Day 7 of the study
  Arms: 1
Other: Placebo — solution, matching placebo to 500 mg PF-00572778, single dose, Days 1 and 7 of the study
  Arms: 2
Drug: PF-00572778 — solution, 500 mg, single dose, only on Day 7 of the study
  Arms: 3

SUMMARY:
PF-00572778, a CRH antagonist, is expected to attenuate adrenocorticotropin (ACTH) and cortisol responses to naloxone by blocking the effect of the CRH increases induced by naloxone at the postsynaptic receptors. Demonstration of a statistically significant attenuation of naloxone induced increases in cortisol and/or ACTH concentrations by PF-00572778 compared to placebo would thus constitute proof of mechanism for the compound. Therefore, this study is to evaluate pharmacodynamic effects of PF-00572778 following naloxone challenge in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and/or female subjects between the ages of 18 and 45 years; Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease; Family (1st degree relatives) and personal history of meeting Diagnostic and Statistical Manual -IV (DSM-IV) criteria for alcohol abuse or dependence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-09; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Area under the cortisol concentration time curve from 0 to 3 hours ( AUC(0-3) ) following naloxone challenge | 1st day on treatment

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | 1st day on treatment
Time to reach the maximum observed serum concentration (Tmax) | 1st day on treatment
Safety laboratory tests, vital signs, ECGs, adverse events monitoring, and physical<br>examinations | 34 days (weekly)
Peak concentrations for plasma cortisol and ACTH | 1st day on treatment
Area under the concentration-time curve from time = 0 to time of the last quantifiable serum PF-00572778 concentration (AUClast) | 2nd day on treatment (Days 6-7)
Area under the ACTH concentration curve from 0 to 3 hours ( AUC(0-3) ) following naloxone challenge | 1st day on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States